CLINICAL TRIAL: NCT03914456
Title: Assessment of Functional Neurorehabilitation in Spinal Cord Injury Using Fmri and Other Neuroimage Tools.
Brief Title: Assessment of Neurorehabilitation in Spinal Cord Injury Using Neuroimage Tools.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/3639
Record Dates: First submitted 2019-03-29; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2007-02

CONDITIONS: Injuries, Spinal Cord
Keywords: Spinal Cord Injury; Motor rehabilitation; Sensorimotor reorganization; Robotic; Functional magnetic resonance imaging
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Seven SCI patients with ASIA C and D participated in this study. They were submitted to a motor-task functional magnetic resonance imaging study (fMRI) before and after the rehabilitation treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body Weight Supported Treadmill Training (Experimental): The rehabilitation program consisted of five hours per day of the treatment, five times a week for two months (40 sessions). The treatment protocol included kinesiotherapy (passive and active mobilizations, muscle lengthening), BWSTT, bicycle, manual therapy (with and without assistance of a mechanical device) and daily life activities training. The duration of each event was approximately one hour.
  The initial time of the treatment on the BWSTT was 20 minutes, and the modification of the time depended on the endurance and capability of each patient. Training charge began at 40% body weight supported and at treadmill speeds of at least 1.5 km per hour. The treadmill speed was increased progressively to 2.5 km per hour, and the level of weight supported was adjusted within sessions to achieve knee extension.
  Interventions: Other: rehabilitation treatment

INTERVENTIONS:
Other: rehabilitation treatment

SUMMARY:
The sensorimotor cortex may play a role in the functional recovery after Spinal Cord Injury (SCI) through efference generated in the absence of the afference. OBJECTIVE: The purpose of this study was to evaluate the potential reorganization in the sensorimotor cortex in SCI patients after Body Weight Supported Treadmill Training (BWSTT) associated with conventional motor rehabilitation. METHOD: Seven SCI patients with ASIA C and D participated in this study. They were submitted to a motor-task functional magnetic resonance imaging study (fMRI) before and after the rehabilitation treatment.

DETAILED DESCRIPTION:
Motor Rehabilitation The rehabilitation program consisted of five hours per day of the treatment, five times a week for two months (40 sessions). The treatment protocol included kinesiotherapy (passive and active mobilizations, muscle lengthening), BWSTT, bicycle, manual therapy (with and without assistance of a mechanical device) and daily life activities training. The duration of each event was approximately one hour.

The initial time of the treatment on the BWSTT was 20 minutes, and the modification of the time depended on the endurance and capability of each patient. Training charge began at 40% body weight supported and at treadmill speeds of at least 1.5 km per hour. The treadmill speed was increased progressively to 2.5 km per hour, and the level of weight supported was adjusted within sessions to achieve knee extension. Table 1 shows the initial and final training parameters for each patient.

To assess functional ability, each patient was assigned a Walking Index for Spinal Cord Injury (WISCI II) (Ditunno and Ditunno 2001) (Table 1), Manual Muscle Testing and Functional Independence Measure (FIM) before and after the treatment period (Table 2).

fMRI Protocol The patients were scanned using a 3T Siemens TIM TRIO system before and after the rehabilitation treatment protocol. The fMRI protocol consisted of a two motor-task fMRI series with the following technical parameters: TE=29 ms; TR=2000 ms, number of slices=36, matrix=128x128, FOV=240 mm, slice thickness= 3 mm; and FA=90º. The patients were given instructions for the motor task they were to perform prior to each scan. The patients were positioned with comfortable pads below the knee to allow the active movement of the ankle. During the functional imaging, each motor activation period was signalled with a short instruction to the subject through the headphones.

The motor task for the fMRI exploration of the foot was the ankle plantar flexion and toe flexion. The block design began with a 20 second rest period, followed by 30 second periods of movement of the right foot, 30 seconds of the left foot movement and 10 seconds of rest. This cycle was repeated three times. The movement performance was controlled visually by two examiners to monitor any movement or apparent change during the rest periods of the non-moving limbs. The patients were oriented to perform the motor task through a voluntary movement. Approximately 15 repetitions were made in each period.

Finally, a T1-weighted structural image of the whole brain was acquired to a perfect localization of activation areas. Acquisition parameters of the structural image were TE= 2.98 ms; TR= 2300 ms; T1= 900 ms; matrix= 256x256; FA= 9º; and T voxel=1x1x1 m3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASIA C or D (Table 1) and the ability to cooperate with instructions of the motor task required. The motor task was to perform ankle plantar flexion, toe flexion and fingers and thumbs movement of both sides; they also had to be able to fulfill the general conditions necessary for an MRI exploration.

Exclusion Criteria:

* Patients with uncontrollable spasticity-induced body movements.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-02-02 (Actual); Primary Completion 2007-09-02 (Actual); Study Completion 2007-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in blood oxygen level (BOLD) signal after motor rehabilitation, evaluated by functional magnetic resonance imaging study (fMRI) | 2 hour
  The blood oxygen level (BOLD) signal in the sensorimotor area, before and after motor rehabilitation, was evaluated by functional magnetic resonance imaging study (fMRI). The signals were obtained through the motor task of the foot: ankle plantar flexion and toe flexion. The block design began with a 20 second rest period, followed by 30 second periods of movement of the right foot, 30 seconds of the left foot movement and 10 seconds of rest. This cycle was repeated three times.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucareli PR, Lima MO, Lima FP, de Almeida JG, Brech GC, D'Andrea Greve JM. Gait analysis following treadmill training with body weight support versus conventional physical therapy: a prospective randomized controlled single blind study. Spinal Cord. 2011 Sep;49(9):1001-7. doi: 10.1038/sc.2011.37. Epub 2011 May 3. PMID 21537338
- [Background] Winchester P, McColl R, Querry R, Foreman N, Mosby J, Tansey K, Williamson J. Changes in supraspinal activation patterns following robotic locomotor therapy in motor-incomplete spinal cord injury. Neurorehabil Neural Repair. 2005 Dec;19(4):313-24. doi: 10.1177/1545968305281515. PMID 16263963